CLINICAL TRIAL: NCT06408376
Title: Physiological Umbilical Cord Clamping in Patients With Congenital Diaphragmatic Hernia. Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital JP Garrahan (Other Government)
Responsible Party: Principal Investigator, Mariela Jozefkowicz, Principal Investigator, Hospital JP Garrahan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1362; 6721 (Other: PRIISA BA)
Record Dates: First submitted 2024-01-22; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Umbilical Cord Clamping; Congenital Diaphragmatic Hernia; Delayed Umbilical Cord Separation
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiological umbilical cord clamping (Experimental): Immediately after birth, the newborn will be placed on a mobile table, made to receive these patients in the delivery room, at the level of the mother's womb, leaving the umbilical cord intact and will be intubated. The patient will be gently ventilated (PIM 15/25 - PEEP 4 - Fio2 50%), until saturation >85% and HR>100 or 10 timed minutes have elapsed, whichever occurs first, the umbilical cord will be clamped and the procedures continued usual reception steps according to the unit´s CDH reception protocol.
  Interventions: Procedure: Physiological cord clamping
- usual reception (No Intervention): Immediately after birth, the newborn is placed on a mobile table, made to receive these patients in the delivery room, at the level of the mother's womb, leaving the umbilical cord intact will be intubated. According to the unit´s CDH reception protocol, patients with CDH cord clamping is done post intubation

INTERVENTIONS:
Procedure: Physiological cord clamping — Immediately after birth, the newborn with prenatal diagnosis of CDH will be placed on a mobile table, made to receive these patients in the delivery room, at the level of the mother's womb, leaving the umbilical cord intact and intubated. The patient will be gently ventilated (PIM 15/25 - PEEP 4 - Fio2 50%), until saturation >85% and HR>100 or 10 timed minutes have elapsed, whichever occurs first, the umbilical cord will be clamped.
  Arms: physiological umbilical cord clamping

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a malformation that affects 1 in every 3000 newborns. The diaphragm does not complete its closure during embryogenesis, which allows the abdominal organs to herniate into the thoracic cavity altering lung development. The lungs of patients with CDH are small, with a decreased surface area for gas exchange and developmental impair of the pulmonary vasculature, resulting in respiratory failure and pulmonary hypertension shortly after birth. When clamping the umbilical cord, a large part of the preload is abruptly excluded, generating an increase in vascular resistance, which in turn increase the afterload, resulting in a decrease in cardiac output. The output is restored by decreasing vascular resistance in pulmonary circuit after lung aeration upon receiving the preload of the right atrium, increasing pulmonary flow and thus sustaining the preload of the left ventricle. If pulmonary aeration occurs before clamping the umbilical cord, the pulmonary blood flow increases before placenta flow is lost, thus avoiding a decrease in cardiac output. This modality has been called physiological base cord clamping (PFC). The hypothesis is that PFC once ventilation has been established could prevent hypoxia and improve cardiac output in newborns with CDH and secondarily improve their hemodynamic parameters, stabilizing gas exchange and pulmonary hypertension during the first 24 hours of birth.

DETAILED DESCRIPTION:
* Type of study: Randomized clinical trial
* Primary objective: To establish the effectiveness of PFC in reducing hypoxia and improving cardiac output compared to immediate postintubation clamping in newborns with CDH. To establish the safety and feasibility of PFC after pulmonary recruitment achieved post intubation.
* Secondary objectives: describe the evolution of patients with CDH 24 hours after birth under pre-established conditions. Relate prenatal indices to the subsequent evolution of these patients. Describe maternal evolution and postpartum complications.
* Population: Patients who attend the Fetal Diagnosis and Treatment program of Garrahan Children's Hospital and undergo prenatal diagnosis of CDH are possible candidates. The study will be carried out in the Neonatal Intensive Care Unit of said hospital.
* Scope of the study: Garrahan Children's Hospital is a level 3 B pediatric hospital and national referral center located in Autonomous City of Buenos Aires, Argentina. Center that receives neonates with CDH referred from all over the country as well as from other countries in the region and carries out the relevant training for equal reception.
* Block randomization: will be carried out on the same day, 2 hours before entering the delivery room
* Intervention: Immediately after birth, the newborn will be placed on a mobile table, made to received these patients in the delivery room, at the level of the mother's womb, leaving the umbilical cord intact, intubated and gently ventilated (positive inspiration pressure (PIM) 15/25 - positive end expiratory pressure (PEEP)4 - fraction of inspired oxygen inspired oxygen fraction (FiO2) 50%), until saturation >85% and heart rate (HR) >100 or 10 timed minutes pass, whichever occurs first, the umbilical cord will be clamped and continued with the usual reception steps in accordance with the unit´s CDH reception protocol.
* Sample size: To calculate the sample size, a prevalence of hemodynamic alterations of 60% was considered in the first 24 hours of life of patients with CDH, following unit statistics and the aforementioned bibliography. The estimated sample size with a relative reduction of 50%: reduction from 60% to 30% of hemodynamic alterations - Power of 80% - Two-tailed test - alpha 5%. 40 patients required in each branch.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal diagnosis of congenital diaphragmatic hernia
* gestational age >34 weeks
* Informed consent signed by the patient's parents

Exclusion Criteria:

* Multiple gestation
* Major malformation or fetal genetic anomaly diagnosed in the prenatal stage
* Emergency cesarean section or maternal condition that prevents the approach
* Lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic deterioration in the first 24 hours of life | 24 hours of life
  Hemodynamic deterioration in the first 24 hours of life (meeting 3 of 4 of the following criteria or entry to extracorporeal membrane oxygenation (ECMO) or Death).
  1. Pre/post ductal saturation difference >10%
  2. Oxygenation index (IO) >20
  3. mean arterial pressure < Percentile 50 or inotrope requirement
  4. Lactic acid >3 mmol/l
complete delivery according group | delivery
  Complete the protocol in the delivery room pre-established according to randomization (yes/no)

SECONDARY OUTCOMES:
Gestational age at diagnosis | 1st day of life
  Gestational age at diagnosis of CDH in weeks
Lung heart rate index observed/expected LHR O/E | from 26 to 32 weeks of gestational age
  lung heart rate index observed/expected (LHR O/E)
liver in thorax | from 26 to 32 weeks of gestational age
  liver in thorax (yes/no) and %
stomach herniation | from 26 to 32 weeks of gestational age
  stomach herniation (yes/no) and %
lung volumen | from 26 to 32 weeks of gestational age
  lung volumen in RMI
Mcgoon | from 26 to 32 weeks of gestational age
  Mcgoon Index in fetal echocardiogram
maternal hematocrit | 1 day before delivery
  maternal hematocrit in gr/dl
Intubation time | From delivery to intubation
  Time to intubation (minutes, seconds)
Cord clamping time | from delivery to cord clamping
  Cord clamping time (minutes, seconds)
Advance resuscitation need on delivery room | from delivery to 30 minutes of life
  Requirement for advanced resuscitation (yes/no) (compressions, drugs, hypothermia)
Time to reach heart rate (HR) >100 | from delivery to 30 minutes of life
  Time to reach HR >100 (minutes, seconds)
Time to reach saturation (SAT) >85% | from delivery to 30 minutes of life
  Time to reach SAT >85% (minutes, seconds)
Cord PH value | inmediatly after cord clampping
  cord ph value
Cord lactic acid value | inmediatly after cord clampping
  cord lactic acid value in mmol/l
saturation at 10 minutes | 10 minutes of life
  pre and post ductal saturation %
Arterial pressure at 10 minutes | 10 minutes of life
  mean arterial tension in mmhg
placenta abruption | 30 minutes of life
  Time for placental abruption (minutes, seconds)
Mother arterial tension after delivery | 10 minutes after delivery
  mothers arterial mean tension after delivery in mmhg
Uterotonic use | 30 minutes after delivery
  uterotonics use on mothers after delivery (yes/no)
Evolution of patient Blood preassure (BP) | 2 - 4 hours and 24 hours of life
  Blood pressure in mmhg
Evolution of patient inotropes required | 2 - 4 hours and 24 hours of life
  Inotrope requirement (yes/no)
Inhaled nitric oxide (NOi) requirement | 2 - 4 hours and 24 hours of life
  NOi requirement (yes/no)
ventilation requirements on the first day | 2 - 4 hours and 24 hours of life
  Ventilatory mode / mean airway pressure (MAP)/ FIo2 %
Oxygenation on the first day | 2 - 4 hours and 24 hours of life
  Partial arterial pressure of oxygen (PaO2) mmhg
Oxygenation index (OI) on the first day | 2 - 4 hours and 24 hours of life
  OI
near-infrared spectroscopy (Nirs) on the first day | 2 - 4 hours and 24 hours of life
  Cerebral and somatic NIRS
B natriuretic peptide (BNP) on the first day | 24 hours of life
  B natriuretic peptide (BNP)
PH value on the first day | 6 and 24 hours of life
  echocardiographic pulmonary hypertension PH (<50% of systemic pressure, between 50-80% of systemic pressure, between 80 and 100% of systemic pressure, systemic, suprasystemic)
cardiac malformations | 6 hours of life
  cardiac malformation (yes/no)
Mortality | through study completion, an average of 1 year
  Mortality (yes/no)
Admission to ECMO | through study completion, an average of 1 year
  Admission to ECMO after the first 24 hours (yes/no)

OTHER OUTCOMES:
maternal age | through study completion, an average of 1 year
  maternal age during pregnancy
maternal history | through study completion, an average of 1 year
  maternal pathological history during pregnancy (yes/no)
baby weight | 30 minutes of life
  Weight in grams
Patent ductus arteriosus (PAD) on the first day (size) | 6 and 24 hours of life
  Patent ductus arteriosus (PAD): size in milimeters
Patent ductus arteriosus (PAD) on the first day (gradient) | 6 and 24 hours of life
  Patent ductus arteriosus (PAD): gradient
Patent ductus arteriosus (PAD) on the first day (shunt direction) | 6 and 24 hours of life
  Patent ductus arteriosus (PAD): shunt direction
Patent foramen ovale (PFO) on the first day (shunt direction) | 6 and 24 hours of life
  Patent foramen ovale (PFO): shunt direction.
Right ventricle (RV) on the first day diameter | 6 and 24 hours of life
  Right ventricle (RV): RV diameter in milimeters
Right ventricle (RV) on the first day TAPSE | 6 and 24 hours of life
  Right ventricle (RV): TAPSE
Tricuspide Insufitienty | 6 and 24 hours of life
  tricuspide insufitienty
Right ventricle funtion | 6 and 24 hours of life
  Right ventricle global disfuntion : no, mild, moderate or severe
Left ventricle (LV) on the first day (eccentricity index) | 6 and 24 hours of life
  Left ventricle (LV): eccentricity index
Left ventricle (LV) on the first day (ejection fraction) | 6 and 24 hours of life
  Left ventricle (LV): ejection fraction (EF)
Left ventricle (LV) on the first day global funtion | 6 and 24 hours of life
  Left ventricle (LV) global disfuntion : no, global disfuntion : no, mild, moderate or severe
Interventricular septum (IS) on the first day | 6 and 24 hours of life
  Interventricular septum: configuration
Pulmonary hypertation grade on the first day | 6 and 24 hours of life
  Pulmonary hypertation: no, mild, moderate or severe
Associated malformations | 24 hours of life
  Associated malformations (yes/no), which
Chromosomopathy or genetic alteration | through study completion, an average of 1 year
  Chromosomopathy or genetic alteration (yes/no), which
Hyperbilirubinemia | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Hyperbilirubinemia requiring phototherapy or exchange transfusion (yes/no)
Early sepsis | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Early sepsis (yes/no)
Omphalitis | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Omphalitis (yes/no)
CDH surgery | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  CDH surgery (yes/no), days of life
Surgical classification | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Surgical classification of CDH (a-b-c-d)
Days in neonatal intensive care unit (NICU) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Days in NICU

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Jozefkowicz, Principal Investigator — Hospital JP Garrahan
Locations (1):
- Hospital de Pediatría S.A.M.I.C. "Prof. Dr. Juan P. Garrahan", Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langham MR Jr, Kays DW, Ledbetter DJ, Frentzen B, Sanford LL, Richards DS. Congenital diaphragmatic hernia. Epidemiology and outcome. Clin Perinatol. 1996 Dec;23(4):671-88. PMID 8982563
- [Background] Keller RL. Antenatal and postnatal lung and vascular anatomic and functional studies in congenital diaphragmatic hernia: implications for clinical management. Am J Med Genet C Semin Med Genet. 2007 May 15;145C(2):184-200. doi: 10.1002/ajmg.c.30130. PMID 17436304
- [Background] Snoek KG, Reiss IK, Greenough A, Capolupo I, Urlesberger B, Wessel L, Storme L, Deprest J, Schaible T, van Heijst A, Tibboel D; CDH EURO Consortium. Standardized Postnatal Management of Infants with Congenital Diaphragmatic Hernia in Europe: The CDH EURO Consortium Consensus - 2015 Update. Neonatology. 2016;110(1):66-74. doi: 10.1159/000444210. Epub 2016 Apr 15. PMID 27077664
- [Background] Bhatt S, Alison BJ, Wallace EM, Crossley KJ, Gill AW, Kluckow M, te Pas AB, Morley CJ, Polglase GR, Hooper SB. Delaying cord clamping until ventilation onset improves cardiovascular function at birth in preterm lambs. J Physiol. 2013 Apr 15;591(8):2113-26. doi: 10.1113/jphysiol.2012.250084. Epub 2013 Feb 11. PMID 23401615
- [Background] Polglase GR, Dawson JA, Kluckow M, Gill AW, Davis PG, Te Pas AB, Crossley KJ, McDougall A, Wallace EM, Hooper SB. Ventilation onset prior to umbilical cord clamping (physiological-based cord clamping) improves systemic and cerebral oxygenation in preterm lambs. PLoS One. 2015 Feb 17;10(2):e0117504. doi: 10.1371/journal.pone.0117504. eCollection 2015. PMID 25689406
- [Background] Hooper SB, Te Pas AB, Lang J, van Vonderen JJ, Roehr CC, Kluckow M, Gill AW, Wallace EM, Polglase GR. Cardiovascular transition at birth: a physiological sequence. Pediatr Res. 2015 May;77(5):608-14. doi: 10.1038/pr.2015.21. Epub 2015 Feb 4. PMID 25671807
- [Background] Horn-Oudshoorn EJJ, Knol R, Te Pas AB, Hooper SB, Cochius-den Otter SCM, Wijnen RMH, Schaible T, Reiss IKM, DeKoninck PLJ. Perinatal stabilisation of infants born with congenital diaphragmatic hernia: a review of current concepts. Arch Dis Child Fetal Neonatal Ed. 2020 Jul;105(4):449-454. doi: 10.1136/archdischild-2019-318606. Epub 2020 Mar 13. PMID 32170029
- [Background] Hooper SB, Polglase GR, te Pas AB. A physiological approach to the timing of umbilical cord clamping at birth. Arch Dis Child Fetal Neonatal Ed. 2015 Jul;100(4):F355-60. doi: 10.1136/archdischild-2013-305703. Epub 2014 Dec 24. PMID 25540147
- [Background] Lefebvre C, Rakza T, Weslinck N, Vaast P, Houfflin-Debarge V, Mur S, Storme L; French CDH Study Group. Feasibility and safety of intact cord resuscitation in newborn infants with congenital diaphragmatic hernia (CDH). Resuscitation. 2017 Nov;120:20-25. doi: 10.1016/j.resuscitation.2017.08.233. Epub 2017 Aug 30. PMID 28860014
- [Background] Duley L, Dorling J, Pushpa-Rajah A, Oddie SJ, Yoxall CW, Schoonakker B, Bradshaw L, Mitchell EJ, Fawke JA; Cord Pilot Trial Collaborative Group. Randomised trial of cord clamping and initial stabilisation at very preterm birth. Arch Dis Child Fetal Neonatal Ed. 2018 Jan;103(1):F6-F14. doi: 10.1136/archdischild-2016-312567. Epub 2017 Sep 18. PMID 28923985
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] Rabe H, Gyte GM, Diaz-Rossello JL, Duley L. Effect of timing of umbilical cord clamping and other strategies to influence placental transfusion at preterm birth on maternal and infant outcomes. Cochrane Database Syst Rev. 2019 Sep 17;9(9):CD003248. doi: 10.1002/14651858.CD003248.pub4. PMID 31529790
- [Background] Katheria AC, Brown MK, Faksh A, Hassen KO, Rich W, Lazarus D, Steen J, Daneshmand SS, Finer NN. Delayed Cord Clamping in Newborns Born at Term at Risk for Resuscitation: A Feasibility Randomized Clinical Trial. J Pediatr. 2017 Aug;187:313-317.e1. doi: 10.1016/j.jpeds.2017.04.033. Epub 2017 May 16. PMID 28526223
- [Background] McGillick EV, Davies IM, Hooper SB, Kerr LT, Thio M, DeKoninck P, Yamaoka S, Hodges R, Rodgers KA, Zahra VA, Moxham AM, Kashyap AJ, Crossley KJ. Effect of lung hypoplasia on the cardiorespiratory transition in newborn lambs. J Appl Physiol (1985). 2019 Aug 1;127(2):568-578. doi: 10.1152/japplphysiol.00760.2018. Epub 2019 Jun 13. PMID 31194603
- [Background] Kashyap AJ, Hodges RJ, Thio M, Rodgers KA, Amberg BJ, McGillick EV, Hooper SB, Crossley KJ, DeKoninck PLJ. Physiologically based cord clamping improves cardiopulmonary haemodynamics in lambs with a diaphragmatic hernia. Arch Dis Child Fetal Neonatal Ed. 2020 Jan;105(1):18-25. doi: 10.1136/archdischild-2019-316906. Epub 2019 May 23. PMID 31123056
- [Background] Sakurai Y, Azarow K, Cutz E, Messineo A, Pearl R, Bohn D. Pulmonary barotrauma in congenital diaphragmatic hernia: a clinicopathological correlation. J Pediatr Surg. 1999 Dec;34(12):1813-7. doi: 10.1016/s0022-3468(99)90319-6. PMID 10626861
- [Background] Foglia EE, Ades A, Hedrick HL, Rintoul N, Munson DA, Moldenhauer J, Gebb J, Serletti B, Chaudhary A, Weinberg DD, Napolitano N, Fraga MV, Ratcliffe SJ. Initiating resuscitation before umbilical cord clamping in infants with congenital diaphragmatic hernia: a pilot feasibility trial. Arch Dis Child Fetal Neonatal Ed. 2020 May;105(3):322-326. doi: 10.1136/archdischild-2019-317477. Epub 2019 Aug 28. PMID 31462406
- [Background] Winter J, Kattwinkel J, Chisholm C, Blackman A, Wilson S, Fairchild K. Ventilation of Preterm Infants during Delayed Cord Clamping (VentFirst): A Pilot Study of Feasibility and Safety. Am J Perinatol. 2017 Jan;34(2):111-116. doi: 10.1055/s-0036-1584521. Epub 2016 Jun 15. PMID 27305177
- [Background] Katheria A, Poeltler D, Durham J, Steen J, Rich W, Arnell K, Maldonado M, Cousins L, Finer N. Neonatal Resuscitation with an Intact Cord: A Randomized Clinical Trial. J Pediatr. 2016 Nov;178:75-80.e3. doi: 10.1016/j.jpeds.2016.07.053. Epub 2016 Aug 26. PMID 27574999
- [Background] Le Duc K, Mur S, Rakza T, Boukhris MR, Rousset C, Vaast P, Westlynk N, Aubry E, Sharma D, Storme L. Efficacy of Intact Cord Resuscitation Compared to Immediate Cord Clamping on Cardiorespiratory Adaptation at Birth in Infants with Isolated Congenital Diaphragmatic Hernia (CHIC). Children (Basel). 2021 Apr 26;8(5):339. doi: 10.3390/children8050339. PMID 33925985